CLINICAL TRIAL: NCT03890822
Title: Coronary Artery Disease Progression in Patients With Acute Coronary Syndromes and Diabetes Mellitus
Acronym: PROGRESSION
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Humanitas Hospital, Italy (Other)
Responsible Party: Principal Investigator, Giulio Stefanini, Head of Clinical Research, Cardio Center, Humanitas Hospital, Italy
Other Study IDs: PROGRESSION
Record Dates: First submitted 2019-03-23; First posted 2019-03-26 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Coronary Artery Disease; Diabetes Mellitus
MeSH Terms: conditions — Coronary Artery Disease; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A total of 100 patients with non-ST-segment elevation acute coronary syndromes with or without diabetes mellitus will be included. All patients will undergo coronary angiography with identification of the infarct-related vessel and percutaneous revascularization with implantation of a stent/scaffold. After revascularization patients will undergo a combined positron emission tomography (PET)-coronary computed tomography (CT) protocol to quantify atherosclerotic burden (i.e. plaque volume) and activity (i.e. 18 fluorum-sodium-fluoride [18FNaF] uptake) in non-infarct related vessels, to assess calcium score (aim 1), and to quantify the acute results of PCI in the infarct-related vessel (aim 2). At 12-month follow-up, all patients will repeat longitudinal 18FNaF PET-coronary CT evaluation to characterize progression of atherosclerosis in the non-infarct related vessels (aim 1) and to quantify neointimal suppression at the site of the treated coronary segment in the infarct-related vessel (aim 2). Blood samples will be collected at baseline and 12 months for all patients.

The aims of the study are:

1. To evaluate coronary artery disease progression in acute coronary syndromes patients with and without diabetes mellitus, and to investigate the predictive value of metabolic profiles, patterns of circulating miRNAs and inflammatory mediators on coronary artery disease progression;
2. To evaluate the progression of disease within the infarct-related vessel treated with the use of bioresorbable stent/bioresorbable polymer stents in diabetic and non-diabetic patients with acute coronary syndromes.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 and <80 years, evidence of non-ST-segment elevation acute coronary syndromes, ability to provide informed consent

Exclusion Criteria:

* ST-segment elevation myocardial infarction, cardiogenic shock, suspected stent thrombosis, known allergy to aspirin or ticagrelor, childbearing potential, life expectancy <1 year due to non-cardiac disease, severe chronic kidney disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with non-ST-segment elevation acute coronary syndrome, with or without diabetes mellitus
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-03-25 (Actual); Primary Completion 2022-03-25 (Estimated); Study Completion 2022-03-25 (Estimated)

PRIMARY OUTCOMES:
Percentual atheroma volume | 12 months
  Assessed by CT
Minimal lumen area | 12 months
  Assessed by CT

SECONDARY OUTCOMES:
Percentual change in 18FNaF uptake | 12 months
Change in minimal lumen area | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Giulio Stefanini, MD, PhD, MSc, Study Chair — Humanitas Research Hospital IRCCS
Locations (1):
- Humanitas Research Hospital, Rozzano, Milan, Italy